CLINICAL TRIAL: NCT01500122
Title: An Open-label, Non Randomized Monocentric Phase I Study Evaluation the Pharmacokinetic Profile of Novel Formulations of RHUDEX®
Brief Title: Study Evaluating the Pharmacokinetic Profile of Novel Formulations of RHUDEX®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CT 5004
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Formulation Finding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: RhuDex — Part 1:
  Regimen A: Rhudex Formulation in Labrafac/ Gelucire Regimen B: Rhudex Formulation in Labrafac/ Aerosil single dose
  The formulation platform (A or B) that shows the best potential to achieve the target PK profile and shows acceptable safety and tolerability will be progressed into part 2 of the study. The purpose of part 2 is to optimize the selected formulation platform. This will be achieved by administrating up to four different formulation compositions.

SUMMARY:
The primary objectives of the study are:

* To compare the pharmacokinetic profiles of RhuDex administered as two novel oral formulations
* To identify the lead formulation and optimise the pharmacokinetic profile by modifying the quantitative composition of that formulation
* Optional: To assess the intravenous pharmacokinetics of RhuDex following administration of an IV microtracer of [14C]RhuDex

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males;
2. Age 18-45 years;
3. Body weight between 70-80 kg;
4. Body Mass Index (BMI) of 18-25 kg/m2;
5. Subject must agree to use an adequate method of contraception (as defined in section 9.4);
6. Must provide written informed consent;
7. Non-smokers (subjects who have never smoked);
8. Absence of cardiovascular risk factors at screening including 12-lead standard ECG, acceptable clinical laboratory tests and the following laboratory parameters within acceptable range: CK; LDH; GPT/GOT (ALAT/ASAT); y-GT, total vs. unconjugated/conjugated serum bilirubin; serum creatinine as judged by the Investigator
9. Must be willing and able to communicate and participate in the whole study.

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months;
2. Subjects who have previously been enrolled in this study;
3. History of any drug or alcohol abuse in the past 2 years;
4. Regular alcohol consumption in males >21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine);
5. A breath carbon monoxide reading of greater than 10 ppm at screening;
6. Radiation exposure from clinical studies, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last twelve months or 10 mSv in the last five years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study;
7. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the Investigator (Section 20);
8. Positive drugs of abuse test result (Section 20);
9. Positive HBV, HCV or HIV results;
10. History of cardiovascular disease,
11. History of sudden death or cardiovascular death before the age of 50 in any first degree relative;
12. History of clinically significant renal, hepatic, respiratory and particularly gastrointestinal disease, especially peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's Disease or Irritable Bowel Syndrome;
13. Any chronic infections e.g. TB
14. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients;
15. Presence or history of allergy requiring treatment. Hayfever is allowed unless it is active;
16. Donation or loss of greater than 400 mL of blood within the previous three months;
17. Subjects receiving prohibited medication as described in Section 9.5;
18. Subjects having received any of the following medication on a regular basis within the previous 3 months: antihypertensives such as ß-blockers, Ca-channel-inhibitors or inhibitors of the renin-angiotensin-system, statins, ASS or any other NSAIDs, diuretics, antacids/PPIs; anticoagulants, antiarrhythmics, antidepressants, antipsychotics;
19. Failure to satisfy the Investigator of fitness to participate for any other reason.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PK blood samples | taken predose, 0.5 h - 1 - 2 - 3 - 4 - 5 - 6 - 7 - 8- 12- 24 -48 - 72 hours after dosing
  All target PK evaluations will be made on the basis that the optimal plasma PK profile will be characterised by a plasma Cmax < 5000 ng/mL, an elimination half-life of > 8h and a C(last) (24h) of around 800-1000 ng/mL. Formulations will explicity not be selected based on determinations of Cmax or AUC(0-inf) alone

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom